CLINICAL TRIAL: NCT00695786
Title: A Phase II Study of Revlimid in Combination With Rituximab as Initial Treatment for Patients With Indolent Non-Hodgkin's Lymphoma (NHL)
Brief Title: Lenalidomide in Combination With Rituximab in Treating Participants With Stage III/IV Indolent Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0042; NCI-2018-01853 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0042 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Ann Arbor Stage III Grade 1 Follicular Lymphoma; Ann Arbor Stage III Grade 2 Follicular Lymphoma; Ann Arbor Stage III Indolent Adult Non-Hodgkin Lymphoma; Ann Arbor Stage III Marginal Zone Lymphoma; Ann Arbor Stage III Small Lymphocytic Lymphoma; Ann Arbor Stage IV Grade 1 Follicular Lymphoma; Ann Arbor Stage IV Grade 2 Follicular Lymphoma; Ann Arbor Stage IV Indolent Adult Non-Hodgkin Lymphoma; Ann Arbor Stage IV Marginal Zone Lymphoma; Ann Arbor Stage IV Small Lymphocytic Lymphoma
MeSH Terms: interventions — Lenalidomide; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Schedule A (lenalidomide, rituximab) (Experimental): Participants receive lenalidomide PO on days 1-21 and rituximab IV over 4-8 hours on day 1 of courses 1-12. Courses repeat every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Lenalidomide; Biological: Rituximab
- Schedule B (lenalidomide, rituximab) (Experimental): Participants receive lenalidomide PO on days 2-22 and rituximab IV over 4-8 hours on days 1, 8, 15, and 22 of course 1 and on day 1 of all subsequent courses. Courses repeat every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Biological: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83

SUMMARY:
This phase II trial studies how well lenalidomide works in combination with rituximab in treating participants with stage III-IV non-Hodgkin lymphoma that is growing slowly. Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth, which may prevent the growth of cancer cells. Monoclonal antibodies, such as rituximab, may interfere with the ability of cancer cells to grow and spread. Giving lenalidomide and rituximab may work better in participants with indolent non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall response rate of lenalidomide in combination with rituximab in previously untreated indolent non-Hodgkin's lymphoma (NHL).

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of lenalidomide in combination with rituximab in previously untreated indolent non-Hodgkin's lymphoma.

OUTLINE: Participants are assigned to 1 of 2 drug schedules.

SCHEDULE A: Participants receive lenalidomide orally (PO) on days 1-21 and rituximab intravenously (IV) over 4-8 hours on day 1 of courses 1-12. Courses repeat every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

SCHEDULE B: Participants receive lenalidomide PO on days 2-22 and rituximab IV over 4-8 hours on days 1, 8, 15, and 22 of course 1 and on day 1 of all subsequent courses. Courses repeat every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age >/= 18 at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Untreated indolent non-Hodgkin's lymphoma stage III-IV including small lymphocytic lymphoma, marginal zone lymphoma, grade 1 or 2 follicular lymphoma. (prior radiation for localized disease allowed).
5. At least one measurable lesion according to the International workshop standardized response criteria for non-Hodgkin's lymphomas (IWG) greater than 1.5cm.
6. ECOG performance status of </= 2 at study entry.
7. Laboratory test results within these ranges: Absolute neutrophil count >/= 1.5 x 10^9/L; Platelet count >/=100 x 10^9/L; Serum creatinine </= 2.0 mg/dL; Total bilirubin </=1.5 mg/dL; AST (SGOT) and ALT (SGPT) </=2 x ULN or </=5 x ULN if hepatic metastases are present.
8. Disease free of prior malignancies for >/= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast, or localized prostate cancer treated with curative intent.
9. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
10. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 -14 days prior to and again within 24 hours of prescribing lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing.
11. Men must agree to use a latex condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy.
12. For patients with bulky disease (tumors >5cm) must be able to take aspirin (81 mg or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females.
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any chemotherapy or experimental therapy within 28 days of enrollment.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concurrent use of other anti-cancer agents or experimental treatments.
9. Known positive for HIV or infectious hepatitis type B or C. (Hepatitis B core antibody can be positive if Hep B surface antigen is negative and no HBV DNA in blood, indicating a cleared infection.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-06-10 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Samaniego, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Fowler NH, Nastoupil LJ, Hagemeister FB, Neelapu SS, Fayad LE, LeBlanc D, Samaniego F, Cheah CY. Characteristics and management of rash following lenalidomide and rituximab in patients with untreated indolent non-Hodgkin lymphoma. Haematologica. 2015 Nov;100(11):e454-7. doi: 10.3324/haematol.2015.131144. Epub 2015 Aug 6. No abstract available. PMID 26250576
- [Derived] Fowler NH, Davis RE, Rawal S, Nastoupil L, Hagemeister FB, McLaughlin P, Kwak LW, Romaguera JE, Fanale MA, Fayad LE, Westin JR, Shah J, Orlowski RZ, Wang M, Turturro F, Oki Y, Claret LC, Feng L, Baladandayuthapani V, Muzzafar T, Tsai KY, Samaniego F, Neelapu SS. Safety and activity of lenalidomide and rituximab in untreated indolent lymphoma: an open-label, phase 2 trial. Lancet Oncol. 2014 Nov;15(12):1311-8. doi: 10.1016/S1470-2045(14)70455-3. Epub 2014 Oct 15. PMID 25439689
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from time of protocol activation 06/10/2008 to protocol closure to new patient entry 02/04/2013.
Pre-assignment Details: 156 patients were enrolled to participant: 2 patients were deemed histologically ineligible, 79 patients had follicular lymphoma, 31 patients had marginal zone lymphoma, and 44 patients had small lymphocytic lymphoma.
Groups:
- Other Histology: Other Histology
- Follicular Lymphoma: Follicular Lymphoma
- Marginal Zone Lymphoma: Marginal Zone Lymphoma
- Small Lymphocytic Lymphoma: Small Lymphocytic Lymphoma
Period: Overall Study
Arm/Group | Other Histology | Follicular Lymphoma | Marginal Zone Lymphoma | Small Lymphocytic Lymphoma
Started | 2 | 79 | 31 | 44
Completed | 1 | 67 | 23 | 36
Not Completed | 1 | 12 | 8 | 8
Not completed — Adverse Event | 0 | 3 | 4 | 2
Not completed — Lost to Follow-up | 0 | 5 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 3 | 1
Not completed — Deemed Ineligible | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Other Histology | Follicular Lymphoma | Marginal Zone Lymphoma | Small Lymphocytic Lymphoma | Total
Number analyzed (Participants) | 2 | 79 | 31 | 44 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 62 | 24 | 36 | 123
  >=65 years | 1 | 17 | 7 | 8 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 39 | 18 | 18 | 75
  Male | 2 | 40 | 13 | 26 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 6 | 4 | 14
  Not Hispanic or Latino | 2 | 54 | 20 | 30 | 106
  Unknown or Not Reported | 0 | 21 | 5 | 10 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 4 | 6
  White | 2 | 72 | 23 | 35 | 132
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 5 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 2 | 77 | 31 | 44 | 154
  United Arab Emirates | 0 | 2 | 0 | 0 | 2
Lymphoma - Non-Hodgkin Stages [Count of Participants; unit: Participants] — Staging at the time of this protocol enrollment included the assessment of certain symptoms to help describe the disease. Stage I cancers are less advanced and often have a better prognosis (outlook). Higher stage cancers typically have spread farther (or have other concerning features), so they might require more intense (or different kinds of) treatment.
  Participants
    Stage I | 0 | 0 | 1 | 0 | 1
    Stage III | 0 | 35 | 9 | 2 | 46
    Stage IV | 2 | 44 | 21 | 42 | 109
Bone Marrow Involvement (+) [Count of Participants; unit: Participants] | 2 | 35 | 9 | 2 | 48
Splenomegaly (+) [Count of Participants; unit: Participants] | 1 | 6 | 5 | 7 | 19
Participants with B Symptoms (+) [Count of Participants; unit: Participants] — Patient experienced the following symptoms unexplained weight loss of more than 10% of their original body weight during the 6 months before diagnosis, unexplained fever with temperatures above 100.4ºF (38ºC), drenching night sweats. Most patients say that either their nightclothes or the sheets on the bed are actually soaked. Sometimes, heavy sweating occurs during the day.
  Participants | 1 | 10 | 3 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Overall Disease Response
Description: Will be monitored simultaneously for each of the subgroups separately using the Bayesian approach of Thall, Simon, Estey. Summary statistics will be provided for continuous variables. Frequency tables will be used to summarize categorical variables. Logistic regression will be will be utilized to assess the effect of patient prognostic factors on the response rate.
Time Frame: At the end of 3 courses (84 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Other Histology | Follicular Lymphoma | Marginal Zone Lymphoma | Small Lymphocytic Lymphoma
Number analyzed (Participants) | 2 | 79 | 31 | 44
Participants
  Best Overall Response - CR | 0 | 56 | 17 | 8
  Best Overall Response - CRu Response | 0 | 13 | 2 | 5
  Best Overall Response - PR | 1 | 6 | 4 | 21
  Best Overall Response - SD | 0 | 1 | 3 | 3
  Best Overall Response - PD | 0 | 0 | 1 | 6
  Best Overall Response - Inevaluable | 1 | 3 | 4 | 1

ADVERSE EVENTS:
Time Frame: beginning at the start of intervention and through 30 days post intervention completion, up to 366 days
Arm/Group | Other Histology | Follicular Lymphoma | Marginal Zone Lymphoma | Small Lymphocytic Lymphoma
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/79 | 0/31 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/2 | 8/79 | 4/31 | 12/44
Other Adverse Events (participants affected / at risk) | 0/2 | 0/79 | 0/31 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Other Histology (N=2) | Follicular Lymphoma (N=79) | Marginal Zone Lymphoma (N=31) | Small Lymphocytic Lymphoma (N=44)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cytokine Release (General disorders) | 1 | 1 | 1 | 0
Cardiac General (Other) (Cardiac disorders) | 0 | 2 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Ischemia cardiovascular (Nervous system disorders) | 0 | 0 | 0 | 1
Memory Loss (Nervous system disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary (Other) (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 8 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT00695786/Prot_SAP_000.pdf